CLINICAL TRIAL: NCT01878266
Title: Prospective Randomized Trial of Two Hypofractionated Radiotherapy Regimens Versus Conventional Radiotherapy in Pediatric Diffuse Brainstem Glioma
Brief Title: Prospective Trial of Two Hypofractionated Radiotherapy Regimens Versus Conventional Radiotherapy in Diffuse Brainstem Glioma in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Cancer Hospital Egypt 57357 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCHE-BT002
Record Dates: First submitted 2013-06-09; First posted 2013-06-14 (Estimated); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Pediatric Brain Stem Glioma
Keywords: Diffuse Intrinsic Pontine Glioma (DIPG); Hypofractionated Radiotherapy; Radiotherapy; Median survival
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hypofractionated Arm (1) (Experimental): A total dose of 39 Gy in daily fractions of 3 Gy, 5 Fractions per week , by conformal radiotherapy sparing of the supratentorial brain. The planning target volume included the tumor as defined by the T2-weighted MRI images with a margin of 1.5-2.0 cm. Margins were adjusted for bony structures and tentorium. With exception of steroids, no neoadjuvant, concomitant, or adjuvant systemic treatment was allowed
  Interventions: Radiation: Hypofractionated Arm (1)
- Hypofractionated Arm (2) (Experimental): The same planning and treatment procedures will be performed. The total dose will be 4500 cGy in 15 fractions in 3 weeks; giving 300 cGy per fraction.
  Interventions: Radiation: Hypofractionated Arm (2)
- Conventional Arm (3) (Other): The same planning and treatment procedures will be performed with 54.0 Gy in 30 fractions giving 1.8 Gy per fraction.
  Interventions: Radiation: Conventional Arm (3)

INTERVENTIONS:
Radiation: Hypofractionated Arm (1) — A total dose of 39 Gy in daily fractions of 3 Gy, 5 Fractions per week
  Arms: Hypofractionated Arm (1)
Radiation: Hypofractionated Arm (2) — The total dose to 4500 cGy in 15 fractions in 3 weeks
  Arms: Hypofractionated Arm (2)
Radiation: Conventional Arm (3) — A total dose of 54 Gy in 30 fractions giving 1.8 Gy per fraction.Conventional arm
  Arms: Conventional Arm (3)

SUMMARY:
This Trial offers a reduction in patient burden, which is especially preferable in children with a poor compliance and poor performance status. This prospective randomized trial was extension to the previous controlled prospective study performed in Children's Cancer Hospital, Egypt and registered at clinicaltrials.com (NCT01635140). The ultimate aim of this work is to demonstrate noninferiority of the hypofractionated regimens relative to the conventional regimen in a controlled randomized clinical study.

DETAILED DESCRIPTION:
In this study will add a third arm in which we will increase in the total dose to 4500 cGy in 15 fractions in 3 weeks may lead to improvement in Over-all survival or Progression-Free Survival.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed patients with a diffuse intrinsic brainstem glioma
2. Aged 2-18years,
3. Have symptoms for less than 3 months and at least two findings of the neurologic triad: cranial nerve deficits, ataxia, or long tract signs.
4. No performance criteria were required for entry onto the study.

Exclusion Criteria:

* Children were not eligible if they had received any prior therapy other than steroids Treatment

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 119 (Actual)
Dates: Start 2013-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Median overall-free survival | 3 years

SECONDARY OUTCOMES:
Progression-free survival | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Cancer Hospital Egypt 57357, Cairo, Egypt